

# TITLE PAGE

| Document Number: | c06524595-04 |
|---|---|
| BI Study Number: | 1237.45 |
| BI Investigational Product(s): | Spiolto <sup>®</sup> Respimat <sup>®</sup> |
| Title: | Assessment of physical functioning and handling of Spiolto <sup>®</sup> Respirat <sup>®</sup> in patients with chronic obstructive pulmonary disease (COPD) requiring long-acting dual bronchodilation in routine clinical practice |
| Protocol version identifier: | 3.0 |
| Date of last version of protocol: | 21 April 2017 |
| PASS: | No |
| EU PAS register number: | EUPAS12750 |
| Active substance: | R03AL06 Tiotropium bromide + Olodaterol |
| Medicinal product: | Spiolto® Respimat® 2.5 microgram/2.5 microgram, inhalation solution; tiotropium/olodaterol |
| Product reference: | NL/H/3157/001/DC |
| Procedure number: | n.a. |
| Marketing authorisation holder(s): | Market Authorisation Holder: Boehringer Ingelheim International GmbH Binger Straße 173 55216 Ingelheim am Rhein Study initiator: |
| Joint PASS: | No |
| Research question and objectives: | The objective of this NIS is to measure changes in physical functioning – a surrogate for physical activity and exercise capacity – in COPD patients on treatment with Spiolto <sup>®</sup> Respimat <sup>®</sup> in routine daily treatment after approximately 6 |

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| | weeks. |
|---|---|
| | A secondary objective is to evaluate the patient's general condition (physician's evaluation) from Visit 1 (baseline visit at the start of the study) to Visit 2 (final visit at the end of the study, approx. 6 weeks after Visit 1), as well as patient satisfaction with Spiolto <sup>®</sup> Respimat <sup>®</sup> at Visit 2. |
| Country(-ies) of study: | 6 countries: Belgium, Denmark, Sweden, The Netherlands,<br>Luxembourg, Portugal |
| Author: | (Medical Team Respiratory MIDI) |
| | Mobile: (Trial Clinical Monitor) |
| | Mobile: |
| EU PAS Register Number | EUPAS12750 |
| Date: | 21 April 2017 |

**Proprietary confidential information** 

© 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved. This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 1. TABLE OF CONTENTS

| TITL | E PAG | E | 1 |
|------|--------|--------------------------------------------------|----|
| 1. | TABL | E OF CONTENTS | 3 |
| 2. | LIST ( | OF ABBREVIATIONS | 5 |
| 3. | RESPO | ONSIBLE PARTIES | 6 |
| 4. | ABSTI | RACT | 7 |
| 5. | AMEN | IDMENTS AND UPDATES | 10 |
| 6. | MILES | STONES | 12 |
| 7. | RATIO | ONALE AND BACKGROUND | 13 |
| 7.1 | ME | DICAL BACKGROUND | 13 |
| 7.2 | DR | UG PROFILE | 14 |
| 8. | RESEA | ARCH QUESTION AND OBJECTIVES | 15 |
| 8.1 | RA | TIONALE FOR PERFORMING THE STUDY | 15 |
| 8.2 | STU | JDY OBJECTIVES | 15 |
| 9. | RESEA | ARCH METHODS | 16 |
| 9.1 | STU | JDY DESIGN | 16 |
| 9 | .1.1 | Outcomes | 17 |
| 9.2 | SET | TTING | 17 |
| 9 | .2.1 | Selection of Patient Population | |
| 9 | .2.2 | Inclusion criteria | 18 |
| 9 | .2.3 | Exclusion criteria | 18 |
| 9.3 | VA | RIABLES | 19 |
| 9.4 | | TA SOURCES | |
| 9.5 | STU | JDY SIZE | 20 |
| 9.6 | | TA MANAGEMENT | |
| 9.7 | | TA ANALYSIS | |
| | .7.1 | Statistical design – Model | |
| | .7.2 | Null and alternative hypotheses | |
| | .7.3 | Planned analyses | |
| | .7.4 | Handling of missing data | |
| 9.8 | _ | ALITY CONTROL | |
| 9.9 | | MITATIONS OF THE RESEARCH METHODS | |
| 9.10 | | HER ASPECTS | |
| 9 | .10.1 | Informed Consent, Data Protection, Study Records | 43 |

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| | 9.10.1.1 | Study Approval, Patient Information, and Informed Consent | 24 |
|---|---|---|---|
| | 9.10.1.2 | Data Quality Assurance | 24 |
| | 9.10.1.3 | Records | 24 |
| | 9.10.1.3.1 | Source Documents | 25 |
| | 9.10.1.3.2 | Direct Access to Source Data and Documents | 25 |
| | 9.10.1.4 | Statement of Confidentiality | 25 |
| | 9.10.1.5 | Completion of Study | |
| | 9.10.1.6 | Protocol Violations | |
| 10. | PROTECT | ION OF HUMAN SUBJECTS | |
| 11. | | MENT AND REPORTING OF ADVERSE EVENTS/ADVERSE NS | |
| 11. | 1 DEFINI | TIONS OF ADVERSE EVENTS28 | |
| 11.2 | | SE EVENT AND SERIOUS ADVERSE EVENT COLLECTION AND TING | ) |
| 11. | 3 REPOR | TING TO HEALTH AUTHORITIES | |
| 12. | | PR DISSEMINATING AND COMMUNICATING STUDY RESULTS | |
| 13. | REFEREN | CES | |
| 13. | 1 PUBLIS | HED REFERENCES | |
| 13.2 | 2 UNPUB | LISHED REFERENCES | |
| ANN | NEX 1. LIST | OF STAND-ALONE DOCUMENTS | |
| ANN | NEX 2. ENC | EPP CHECKLIST FOR STUDY PROTOCOLS | |
| ANN | NEX 3. ADD | ITIONAL INFORMATION | |

#### BI Study Number 1237.45

c06524595-04

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 2. LIST OF ABBREVIATIONS

ADR Adverse Drug Reaction

AE Adverse Event

BI Boehringer Ingelheim
CA Competent Authority
CI Confidence Interval
CML Local Clinical Monitor

COPD Chronic Obstructive Pulmonary Disease

CRA Clinical Research Associate eCRF Electronic Case Report Form DMP Data Management Plan

EU European Union FDC Fix Dose Combination

FEV1 Forced expiratory volume in one second

GCP Good Clinical Practice

GEP Good Epidemiological Practice

GPP Good Pharmacoepidemiology Practice

GOLD Global Initiative for Chronic Obstructive Lung Disease

ICH International Conference on Harmonisation

ICS Inhalative Corticosteroides
IEC Independent Ethics Committee

ISF Investigator Site File

LABA Long-acting beta<sub>2</sub> adrenoceptor agonist LAMA Long-acting muscarinic antagonist

MedDRA Medical Dictionary for Drug Regulatory Activities

mMRC Modified Medical Research Council

NIS Non-Interventional Study PF-10 Patient questionnaire

PGE Physician's Global Evaluation

SAE Serious Adverse Event SAP Statistical Analysis Plan SD Standard Deviation

SF-36 36-Item Short Form Health Survey
SGRQ St George's Respiratory Questionnaire
SmPC Summary of Product Characteristics

WHO World Health Organisation

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 3. RESPONSIBLE PARTIES

| Therapeutic Area Respiratory Medicine (TA ) | |
|---|---|
| Team Member Medical Affairs (TM MA) | _ |
| Team Member Epidemiology (TM Epi) | _ |
| Global Epidemiology ( GEpi) | _ |
| Therapeutic Area Risk Management (TA RM), and Pharmacovigilance Working Group (PVWG) | |
| GPV Study Coordination | |
| Trial Statistician (TSTAT) | |
| Trial Data Manager (TDM) | |
| Trial Programming | |
| Medical Team Respiratory | - |
| Trial Clinical Monitor (TCM) | - |
| Coordinating Investigator (CI) | not applicable |
| CRO – | |

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 4. ABSTRACT

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished mo<br>product:<br>Spiolto® Respimat® | edicinal | | |
| Name of active ingre<br>R03AL06 | edient: | | |
| Tiotropium bromide | + Olodaterol | | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| 02 Mar 2016 | 1237.45 | 3.0 | 21 Apr 2017 |
| Title of study: | Respimat <sup>®</sup> in par | hysical functioning and handlin<br>tients with chronic obstructive p<br>ng long-acting dual bronchodila | oulmonary disease |
| Rationale and background: | Reduced physical activity resulting in deconditioning and restricted physical functioning is a common problem of patients with moderate to severe COPD. Clinical studies investigating treatment with Spiolto® Respimat® and its single components have shown significant improvements in exercise capacity in patients with COPD. Real-world data on the effects of a fixed-dose combination (LABA+LAMA) therapy with tiotropium and olodaterol administered in a single device, in COPD patients who need treatment with two long-acting bronchodilators, is not available. | | |
| Research question and objectives: | The primary objective of this NIS is to measure changes in physical functioning – a surrogate for physical activity and exercise capacity – in COPD patients on treatment with Spiolto® Respimat® in routine daily treatment after approximately 6 weeks. | | |
| | A secondary objective is to evaluate the patient's general condition (physician's evaluation) from Visit 1 (baseline visit at the start of the study) to Visit 2 (final visit at the end of the study, approx. 6 weeks after Visit 1), as well as patient satisfaction with Spiolto <sup>®</sup> Respimat <sup>®</sup> at Visit 2. | | |
| Study design: | Open-label observational study: 6 countries, including COPD patients receiving treatment with Spiolto <sup>®</sup> Respimat <sup>®</sup> for approximately 6 weeks, which is the average time between two medical consultations. | | |
| Population: | COPD patients requiring a fixed combination therapy of two long-<br>acting bronchodilators (LAMA + LABA) according to approved<br>SmPC and GOLD guidelines. | | |
| Variables: | <ul> <li>Patient demographics (age, gender, height &amp; weight)</li> <li>Concomitant diseases / Comorbidities</li> <li>Concomitant medication</li> <li>General condition of patient based on Physician's Global</li> </ul> | | |

## Boehringer Ingelheim  BI Study Number 1237.45

**** 

c06524595-04

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Name of company:<br>Boehringer Ingelhein | ı | | |
|---|---|---|---|
| Name of finished medicinal product: Spiolto® Respimat® | | | |
| Name of active ingre<br>R03AL06<br>Tiotropium bromide | | | |
| Protocol date: Study number: | | Version/Revision: | Version/Revision date: |
| 02 Mar 2016 1237.45 | | 3.0 | 21 Apr 2017 |
| | Evaluation (PGE) - Smoking history - Exacerbations - Breathlessness based on mMRC score - Physical Functioning based on PF-10 scores - Patient satisfaction with Spiolto® Respimat® - Safety; ADR (serious and non-serious), fatal AEs, pregnancies - GOLD spirometric classifications (1, 2, 3, 4) - GOLD patient groups (A, B, C, D) | | |

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished mo<br>product:<br>Spiolto <sup>®</sup> Respimat <sup>®</sup> | edicinal | | |
| Name of active ingre<br>R03AL06 | edient: | | |
| Tiotropium bromide | + Olodaterol | | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| 02 Mar 2016 | 1237.45 | 3.0 | 21 Apr 2017 |
| Data sources: | To be completed by the physician: Patient demographics Patient medical files Physician's Global Evaluation (PGE) at Visit 1 and Visit 2 To be completed by the patient at Visit 1: mMRC breathlessness scale To be completed by the patient at Visit 1 and at Visit 2: Physical Functioning Questionnaire (PF-10) To be completed by the patient at Visit 2 only: Patient satisfaction survey | | |
| Study size: | 1200 patients, 225 sites; 6 countries: Belgium, Denmark, Sweden, The Netherlands, Luxembourg, Portugal | | |
| Data analysis: | Primary outcome: "therapeutic success" at Visit 2 (= 10-point increase in the PF-10 score between Visit 1 and Visit 2). Secondary outcomes: - Changes in the PF-10 score from Visit 1 to Visit 2 - General condition of the patient, evaluated by the physician (PGE score) at Visit 1 and Visit 2. - Patient satisfaction with Spiolto® Respimat® at Visit 2. | | |
| Milestones: | Start of data coll<br>End of data colle<br>Final report of st | ection | September 2016<br>March 2018<br>June 2018 |

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 5. AMENDMENTS AND UPDATES

| Protocol | Protocol v3.0, Amendment 2 | | | |
|---|---|---|---|---|
| Number | Date | Section of study protocol | Amendment or update | Reason |
| 1 | 21 Apr 2017 | Front Page, p. 2 | Changing countries of the study | Deleting Norway,<br>Adding Portugal |
| 2 | 21 Apr 2017 | Front Page, p. 2 | Adding protocol author | New Medical Team<br>Leader Respiratory<br>MIDI |
| 3 | 21 Apr 2017 | Front Page, p. 2 | Adding protocol author | New TCM |
| 4 | 21 Apr 2017 | Paragraph 3<br>Responsible<br>parties, p. 6 | Changing Therapeutic Area Head Risk Management (TAH RM), and Pharmacovigilan ce Working Group (PVWG) chairperson | New Therapeutic Area Head Risk Management (TAH RM), and Pharmacovigilance Working Group (PVWG) chairperson |
| 5 | 21 Apr 2017 | Paragraph 3<br>Responsible<br>parties, p. 6 | Changing Trial<br>Data Manager | New Trial Data<br>Manager |
| 6 | 21 Apr 2017 | Paragraph 3<br>Responsible<br>parties, p. 6 | Changing Trial<br>Programming | New Trial<br>Programmer |
| 7 | 21 Apr 2017 | Paragraph 3<br>Responsible<br>parties, p. 6 | Changing<br>Medical Team<br>Leader<br>Respiratory | New Medical Team<br>Leader Respiratory |
| 8 | 21 Apr 2017 | Paragraph 3<br>Responsible<br>parties, p. 6 | Changing TCM name | New TCM |
| 9 | 21 Apr 2017 | Paragraph 4<br>Abstract, p. 9 | Changing study size | Changing number of sites from 250 to 225 |
| 10 | 21 Apr 2017 | Paragraph 4 | Changing study | Deleting Norway, |

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| | | Abstract, p. 9 | size | Adding Portugal |
|---|---|---|---|---|
| 11 | 21 Apr 2017 | Paragraph 4<br>Abstract, p. 9 | Changing<br>Milestones | Updated date of start of data collection |
| 12 | 21 Apr 2017 | Paragraph 4<br>Abstract, p. 9 | Changing<br>Milestones | Updated date of end of data collection |
| 13 | 21 Apr 2017 | Paragraph 4<br>Abstract, p. 9 | Changing<br>Milestones | Updated date of<br>Final report of study<br>results |
| 14 | 21 Apr 2017 | Paragraph 6, p. 12 | Changing<br>Milestones | Updated date of end of data collection |
| 15 | 21 Apr 2017 | Paragraph 6, p. 12 | Changing<br>Milestones | Updated date of<br>Final report of study<br>results |
| 16 | 21 Apr 2017 | Paragraph 9<br>Research<br>Methods, p. 17<br>and p. 18 | Changing setting (9.2) and Selection of Patient Population (9.2.1.) | Changing number of sites from 250 to 225 |
| 17 | 21 Apr 2017 | Paragraph 9<br>Research<br>Methods, p. 17<br>and p. 18 | Changing setting (9.2) and Selection of Patient Population (9.2.1.) | Deleting Norway,<br>Adding Portugal |
| 18 | 21 Apr 2017 | Paragraph 9<br>Research<br>Methods, p. 18 | Change in exclusion criteria (9.2.3.) | Change in exclusion criterion n°2: "previous 6 weeks" instead of "previous 6 months" |
| 19 | 21 Apr 2017 | Paragraph 9<br>Research<br>Methods, p. 18 | Adding note in exclusion criteria (9.2.3.) | Adding note to clarify exclusion criterion n° 2 |

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 6. MILESTONES

| Milestone | Planned Date |
|--------------------------------|----------------|
| Start of data collection | September 2016 |
| End of data collection | March 2018 |
| Final report of study results: | June 2018 |

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7. RATIONALE AND BACKGROUND

#### 7.1 MEDICAL BACKGROUND

COPD is defined as a preventable and treatable disease of the airways, with significant systemic consequences. Inactivity is believed to be crucial to the development of the extrapulmonary effects of the disease like skeletal muscle weakness, osteoporosis and cardiovascular disease. Recent data suggest that patients suffering from COPD with low levels of physical activity have increased risk for hospital admission and have significantly enhanced mortality. Epidemiological data suggest that this may directly or indirectly lead to more rapid decline in lung function [R13-3633].

Physical activity is reduced early in the disease progression, as of GOLD Stage 2 [R13-3633]. More recent evidence from large placebo controlled clinical trials indicates that COPD patients are experiencing a steeper absolute decline in lung function with GOLD 2 airflow limitation than with GOLD 3 and 4 [R15-5015]. All these observations suggest the importance of early optimal treatment of the disease.

Long-acting bronchodilators, such as long-acting muscarinic antagonists (LAMAs), are the cornerstone of maintenance therapy for patients with moderate to very severe chronic obstructive pulmonary disease (COPD) whose symptoms are not adequately controlled by short-acting bronchodilators alone [P13-05794, P14-01052].

An option recommended by GOLD guideline for patients not adequately controlled on a single long-acting bronchodilator is to combine a LAMA with a long-acting  $\beta$ 2-agonist (LABA) [P14-01052]. This has prompted the development of combining LAMA+LABA as fixed-dose combinations [P13-05794]. The rationale for combining bronchodilators with different mechanisms is based on the notion of additive relaxation of airway smooth muscle by direct inhibition of cholinergic activity and functional antagonism of bronchoconstriction through  $\beta$ 2-adrenergic pathways, with the expectation of an increase in the degree of bronchodilation for equivalent or lesser side effects. Several recent studies have provided evidence in support of this increased bronchodilatory effect when LABAs are added to LAMAs.

When long acting beta-agonists (LABA) and long acting muscarinic antagonists (LAMA) with similar or equivalent posologies are combined, the opportunity exists for offering a simpler and more convenient administration regimen with the development of fixed combinations within the same inhaler device. Fixed-dose combinations of a short-acting  $\beta$ 2–agonist (SABA) and a short-acting anticholinergic (SAMA) have been developed and have been shown to be safe, efficacious and convenient for the patient (e.g., Berodual®: Fenoterolhydrobromid + Ipratropiumbromid, Combivent®: salbutamol + ipratropium bromide; [P94-1346]). Olodaterol is a highly selective and nearly full  $\beta$ 2 agonist [P10-07776, P11-07720] that provides 24-h bronchodilation in patients with COPD [P13-11467, P13-14112, P13-11346, P13-11345]. Olodaterol is also associated with symptomatic benefit [P13-11341] and enhanced exercise capacity [P13-14109].

The complementary modes of action of tiotropium and olodaterol have previously been demonstrated in animal models, phase II clinical trials and during the Phase IIIa programs [P10-09337, P14-12073, P13-02357].

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

In the Phase III programs the additional benefits of the tiotropium + olodaterol fixed-dose combination (FDC) over its mono-components has been assessed on lung function, quality of life (St. George's Respiratory Questionnaire -SGRQ), dyspnea (Transition Dyspnea Index-TDI) and exercise endurance time. Another clinically important potential benefit of the tiotropium + olodaterol FDC over the mono components is the impact on exacerbations of COPD.

#### 7.2 DRUG PROFILE

Tiotropium + olodaterol FDC is an aqueous solution of tiotropium and olodaterol contained in a cartridge. It is administered by using the Respimat<sup>®</sup> inhaler. One cartridge is used per inhaler, which is inserted into the device prior to first use. In pivotal clinical trials and for the intended marketed product, the clinical dose consists of two puffs once daily. The Respimat<sup>®</sup> inhaler uses mechanical energy to create a soft mist which is released over a period of approximately 1.5 seconds.

Tiotropium + olodaterol FDC was shown to be safe and well tolerated over 1 year in a moderate to very severe COPD population. The overall incidences of adverse events (AEs), serious adverse event (SAEs), fatal AEs, frequencies for cardiac events and major adverse cardiovascular event in the tiotropium + olodaterol FDC treatment group were similar to the mono-components. The nature and frequency of AEs in general was consistent with the disease under study. There were no results in the clinical development program suggesting the need for absolute contraindications for the combination product [P15-03349].

In conclusion, the clinical trials conducted to date have shown tiotropium + olodaterol FDC to be a safe, well tolerated and efficacious combination therapy according to treatment guidelines in a moderate to very severe COPD patient population [P15-04531, P15-03349]. The observed incremental bronchodilator response for the combination compared to the individual components translated into benefits that were meaningful to the patient, with improvements in several patient centered outcomes. For further information please refer to the SmPC of Spiolto<sup>®</sup> Respimat<sup>®</sup>.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 8. RESEARCH QUESTION AND OBJECTIVES

#### 8.1 RATIONALE FOR PERFORMING THE STUDY

The contribution of physical inactivity to disability in COPD is difficult to distinguish from disease progression; however, it is clear that physical activity is significantly lower in patients with COPD than in healthy controls [R13-3633].

COPD prevents patients from carrying out daily activities due to exercise intolerance, which is often attributed to limited pulmonary ventilation. Physical inactivity may be related to avoidance of exertion as a result of fear of dyspnea. Furthermore, physical inactivity has been associated with skeletal muscle weakness and exercise intolerance [R15-4559, R15-4561].

The loss of physical activity in COPD is also associated with increased mortality. Data from a study of 2386 patients with COPD demonstrated that, following adjustment for relevant confounders, subjects who reported low, moderate or high physical activity had a significantly lower risk of all-cause mortality than those with very low physical activity (p = 0.001) [R15-4564]. Clinical studies of both Spiriva® [P13-04267, P05-09483, P13-14109] and Striverdi® Respimat® in COPD patients have demonstrated significant improvement in exercise capacity [P13-14109].

The benefits of tiotropium + olodaterol FDC have been studied in controlled Phase III programs on exercise endurance, however, data regarding physical activity when treated with Spiolto<sup>®</sup> Respirat<sup>®</sup> is not available from a real world setting.

#### 8.2 STUDY OBJECTIVES

The primary objective of the study is to measure changes in physical functioning - serving as a surrogate for physical activity and exercise capacity - in COPD patients being treated with Spiolto<sup>®</sup> Respirat<sup>®</sup> after approximately 6 weeks in routine clinical practice.

The secondary objectives are to evaluate the patient's general condition (physician's evaluation) at Visit 1 (baseline visit at the start of the study) and at Visit 2 (final visit at the end of the study, approx. 6 weeks after Visit 1), as well as patient satisfaction with Spiolto<sup>®</sup> Respirat<sup>®</sup> at Visit 2.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 9. RESEARCH METHODS

#### 9.1 STUDY DESIGN

This is a self-controlled study design enrolling consented COPD patients who will be treated with Spiolto<sup>®</sup> Respimat<sup>®</sup> according to the approved SmPC.

Patients will be enrolled consecutively and will be followed over an observational period of approx. 6 weeks. Data as listed in <u>Table 9.1:1</u> will be collected.

Table 9.1:1: Visit flow chart and data collection parameters

| Parameter | Visit 1;<br>baseline<br>visit | Visit 2;<br>approx. 6<br>weeks after<br>baseline visit |
|---|---|---|
| Informed Consent | X | |
| Inclusion / Exclusion Criteria | X | |
| Patient demographics (age, gender, height, and weight) | X | |
| Smoking history | X | X |
| Start of COPD | X | |
| Number of exacerbations in the last 12 months | X | |
| Number of exacerbations leading to hospitalization in the last 12 months | X | |
| Past COPD therapies (6 months before Visit 1) | X | |
| COPD related and other relevant concomitant medication | X | X |
| Concomitant diseases / Comorbidities | X | X |
| Respirat® training (yes/no) | X | |
| COPD severity based on GOLD assessment <sup>1</sup> | X | |
| mMRC breathlessness scale, completed by the patient | X | |
| Physical functioning (PF-10) questionnaire, completed by patient | X | X |
| General condition of patient evaluated by Physician's Global Evaluation (PGE) | X | X |
| Adverse Drug Reactions (serious and non-serious), fatal AE, pregnancy | X | X |
| Patient satisfaction with Spiolto® Respimat®, survey completed by the patient | | X |
| Rational for Spiolto® Respimat® treatment discontinuation (if applicable) | | X |
| Continuation or discontinuation of treatment with Spiolto® Respimat® after the study (yes/no) | | X |

<sup>&</sup>lt;sup>1</sup> GOLD patient group (A, B, C or D) will be automatically calculated within the eCRF based on available exacerbation history, mMRC, and GOLD spirometric classification of airflow limitation based on post-bronchodilator FEV<sub>1</sub> if available.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Baseline characteristics of patients being eligible and who gave Informed Consent, but were not treated in the study will also be collected.

#### 9.1.1 Outcomes

#### **Primary outcome:**

The primary outcome is to measure "Therapeutic success" (as a 10-point increase of PF-10) between Visit 1 and Visit 2 using a physical functioning questionnaire, which is a subdomain of the SF-36 patient questionnaire. The PF-10 sub-domain consists of 10 questions evaluating the extent of experienced restrictions while conducting usual activities. Each question of the PF-10 can be answered with "yes, limited a lot", "yes, limited a little", or "No, not limited at all", with a score of 1, 2, or 3. The scores over the 10 questions will be summed, resulting in a value between 10 (a patient answering all questions with "yes, limited a lot") and 30 (a patient answering all questions with "No, not limited at all"). The final sum of the individual scores will be standardized to a range of 0 to 100 using the following formula: 100\*(sum-10)/20.

#### **Secondary outcomes:**

- Changes in the PF-10 score from Visit 1 to Visit 2
- General condition of the patient, evaluated by the physician (PGE score) at Visit 1 and Visit 2.
- Patient satisfaction with Spiolto<sup>®</sup> Respimat<sup>®</sup> at Visit 2.

#### 9.2 SETTING

It is planned that data of approximately 1200 patients from approximately 225 sites in 6 countries will be collected. Site selection will be performed to reflect routine COPD care in the participating countries to secure representativeness of the COPD population. The following countries will participate in this non-interventional study: Belgium, Denmark, Sweden, The Netherlands, Luxembourg and Portugal.

A log of all patients included into the study (i.e. having given informed consent) will be maintained in the ISF at the investigational site irrespective of whether they have been treated or not.

Boehringer Ingelheim reserves the right to discontinue the study overall or at a particular study site at any time for the following reasons:

- 1. Failure to meet expected enrolment goals overall or at a particular study site
- 2. Emergence of any efficacy/safety information that could significantly affect continuation of the study, or any other administrative reasons, i.e. lack of recruitment
- 3. Violation of the protocol, the contract, or applicable laws and regulations for non-interventional studies, which could disturb the appropriate conduct of the NIS

The investigator / the study site will be reimbursed for reasonable expenses incurred in case of study termination (except in case of the third reason).

**BI Study Number 1237.45** 

c06524595-04

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.2.1 Selection of Patient Population

1200 patients with chronic obstructive pulmonary disease (COPD) in whom combination treatment with long-acting bronchodilators is indicated in accordance with the guidelines are to be observed in approx. 225 sites (hospital and non-hospital pulmonary medicine physicians and general practitioners) as part of this NIS. In the six participating countries (Belgium, Denmark, Sweden, The Netherlands, Luxembourg and Portugal), sites in urban as well as rural areas will be included. The nationwide distribution of the participating sites in the six countries and the number of patients enrolled are intended to ensure that the data collected are representative.

Possible contraindications are to be checked prior to treatment with Spiolto<sup>®</sup> Respimat<sup>®</sup>. See also the latest Summaries of Product Characteristics on Spiolto<sup>®</sup> Respimat<sup>®</sup>.

Every physician is to enrol the first consecutive patients he/she chooses to treat with Spiolto<sup>®</sup> Respirat<sup>®</sup>. The inclusion of four to six patients is planned per site.

The decision to treat will be taken independently of participation in this NIS and will be made before participation is considered.

#### 9.2.2 Inclusion criteria

Patients can be included if all of the following criteria are met:

- 1. Written informed consent prior to participation
- 2. Female and male patients  $\geq 40$  years of age
- 3. Patients diagnosed with COPD and requiring long-acting dual bronchodilation (LAMA + LABA) treatment according to approved Spiolto® Respimat® SmPC and COPD GOLD guideline recommendation

#### 9.2.3 Exclusion criteria

- 1. Patients with contraindications according to Spiolto<sup>®</sup> Respirat<sup>®</sup> SmPC
- 2. Patients who have been treated with a LABA/LAMA combination (free and fixed dose) in the previous 6 weeks

#### Note:

- Patients previously treated with LABA or LAMA (with or without ICS) are eligible to be included in the study.
- Patients previously treated with LABA+LAMA or LABA+LAMA+ICS cannot be included in the study, if they received this treatment in the last 6 weeks.
- 3. Patients continuing LABA-iCS treatment should not be additionally treated with Spiolto® Respirat® in order to avoid a double dosing of long-acting beta-agonists
- 4. Patients for whom further follow-up is not possible at the enrolling site during the planned study period of approx. 6 weeks
- 5. Pregnancy and lactation
- 6. Patients currently listed for lung transplantation
- 7. Current participation in any clinical trial or any other non-interventional study of a drug or device

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.3 VARIABLES

During the observational period, the following data will be collected in an eCRF:

- Patient demographics (age, gender, height & weight)
- Concomitant diseases / Comorbidities such as cardiovascular disease, diabetes mellitus, musculoskeletal impairment, renal diseases, liver diseases, osteoporosis, gastroesophageal reflux (GERD), or lung cancer
- COPD related and other relevant concomitant medication such as beta-blockers, beta-agonists, corticosteroids, or proton pump inhibitors
- General condition of patient based on Physician's Global Evaluation (PGE) to assess the general condition of the patient at the beginning and at the end of the study
- Smoking status (current smoker, former smoker, and never smoker) and pack-years
- Reported exacerbations based on medical history in the last 12 months and exacerbations leading to hospitalization in the last 12 months
- Assessment of the severity of breathlessness based on the Modified Medical Research Council Questionnaire (mMRC score)
- Physical Functioning based on PF-10 scores
- Patient satisfaction with Spiolto<sup>®</sup> Respimat<sup>®</sup> to assess the overall satisfaction with Spiolto<sup>®</sup> Respimat<sup>®</sup> as well as specific inhalation from the device and device handling
- Safety Reporting; Adverse Drug Reactions (serious and non-serious), fatal AEs, pregnancies at the beginning and at the end of the study
- GOLD spirometric classifications (1, 2, 3, 4), based on GOLD guidelines
- GOLD patient groups (A, B, C, D), based on GOLD guidelines

\*The PF-10 is a sub-domain of the SF-36 and consists of 10 questions evaluating the extent of experienced restrictions while conducting usual activities. Each question of the PF-10 can be answered with "yes, limited a lot", "yes, limited a little", or "No, not limited at all", with a score of 1, 2, or 3. The scores over the 10 questions will be summed, resulting in a value between 10 (a patient answering all questions with "yes, limited a lot") and 30 (a patient answering all questions with "No, not limited at all"). The final sum of the individual scores will be standardized to a range of 0 to 100 using the following formula: 100\*(sum-10)/20.

#### 9.4 DATA SOURCES

Patient files (paper and/or electronically) of COPD patients as documented by the treating physician in his/her daily practice will be used as data source.

All participating physicians will be obliged to make a note of the patient's participation in the NIS in the patient's original documents.

In the event of possible queries, the participating physician must be able to identify the patient observed.

Medical information on the patient must be communicated and analysed only using the patient number.

As the physical exercise capacity of the COPD patients cannot be measured directly as part of an NIS, the evaluation of general condition by the physician and an extract from the SF-36 quality-of-life questionnaire relating to physical functioning (PF-10) will be documented as surrogate parameters.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The treating physician will use the Physician's Global Evaluation (PGE) to evaluate the general condition of the patient on an 8-point ordinal scale from 1 (very poor) to 8 (excellent). PGE will be completed before and approx. 6 weeks after treatment initiation.

The modified Medical Research Council (mMRC) scale will be used to assess the breathlessness state of the patient before the treatment. The mMRC stage (0 to 4) collected from the patient, as well as the exacerbation history and the post-bronchodilator FEV<sub>1</sub>, will be used to automatically calculate the GOLD patient group (A, B, C, or D) in the eCRF.

The physical functioning (PF-10) questionnaire is a subscale of the validated 36-Item Short Form Health Survey and contains 10 questions about everyday physical activity and functioning. Patients will be asked to complete the PF-10, in order to evaluate their physical functioning before and after treatment with Spiolto<sup>®</sup> Respimat<sup>®</sup>.

A patient satisfaction survey will also be completed at Visit 2, using a 7-point ordinal scale with divisions from very dissatisfied to very satisfied.

#### 9.5 STUDY SIZE

In a previous study, 205.426 with over 1000 patients treated with Spiriva<sup>®</sup> Respimat<sup>®</sup>, therapeutic success (i.e., 10-point increase in the PF-10 score between Visit 1 and Visit 2) was achieved in 61% of the patients.

However, in the present study a lower therapeutic success rate is expected as patients may be already on maintenance treatment at baseline. Assuming a 50% therapeutic success rate and a sample size of 1116 patients, the 95% confidence interval for the therapeutic success rate would be between 47.1% (lower limit) and 52.9% (upper limit).

To account for a 7% drop-out rate, the sample size becomes 1200 patients.

#### 9.6 DATA MANAGEMENT

A data management plan (DMP) will be created to describe all functions, processes, and specifications for data collection, cleaning and validation. The electronic Case Report Forms (eCRFs) will include programmable edits to obtain immediate feedback if data are missing (also negative answers, unknown), out of range, illogical or potentially erroneous. These rules may encompass simple checks such as range validation or presence/absence of data. Concurrent manual data review may be performed based on parameters dictated by the DMP. Ad hoc queries to the sites may be generated and followed up for resolution. A source data quality audit may be initiated to ensure that the data in the database is accurate. Source data verification (SDV) will be performed at sites identified by a risk-based approach as needed.

The database will be housed in a physically and logically secure computer system maintained in accordance with a written security policy. The system will meet the standards of the International Committee on Harmonization guideline E6R1 regarding electronic study data handling. Patient confidentiality will be strictly maintained.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.7 DATA ANALYSIS

**BI Study Number 1237.45** 

#### 9.7.1 Statistical design – Model

Details will be described in the statistical epidemiological analysis plan (SEAP).

### 9.7.2 Null and alternative hypotheses

No formal hypothesis testing will be performed since this is a self-controlled study.

## 9.7.3 Planned analyses

All patients who have received at least one dose of Spiolto<sup>®</sup> Respimat<sup>®</sup> will be included in the analyses; this is the treated set. All analyses will be performed on the treated set (astreated analysis). If patients have missing values for an outcome, those patients will be excluded for that outcome's analysis. For example, if a patient is missing the PF-10 score at Visit 1 and/or Visit 2, that patient will be excluded from the analyses for the primary endpoint of therapeutic success and the secondary endpoint of change in PF-10 from Visit 1 to Visit 2.

The assessment will be carried out using SAS® software. The statistical characteristics presented in the end-of-text tables will be N / mean / SD / min / median / max for continuous variables. Tabulations of relative and absolute frequencies will be presented for categorical variables. Incidence rates and 95% CI will be given when appropriate.

The analyses will relate to the following data:

- Patient demographics (age, gender, height, and weight);
- Comorbidities (main diagnosis and concurrent diagnosis according to MedDRA, version valid as at the time of database closure);
- COPD related and other concomitant medication (according to the WHO classification, version valid at the time of database closure)
- History of smoking
- Exacerbations
- Breathlessness based on mMRC score at Visit 1
- Physical Functioning based on PF-10 scores (therapeutic success at Visit 2); primary outcome
- Changes from Visit 1 to Visit 2 in the PF-10 score; secondary outcome
- Patient satisfaction with Spiolto<sup>®</sup> Respimat<sup>®</sup> at Visit 2 only; secondary outcome
- General condition of the patient: evaluated by the physician (Physician's Global Evaluation (PGE)); secondary outcome
- Adverse Drug Reactions (ADR & SADR), fatal AEs, pregnancies
- GOLD spirometric classification (1,2, 3, 4)
- GOLD patient groups (A, B, C, D)

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Details of treatment with inhaled respiratory agents before the study
- Details of treatment with respiratory agents during the study
- Reasons for ending treatment during the observation period
- Details of treatment continuation / discontinuation

### Main analysis

For the primary outcome, the proportion of patients with therapeutic success will be presented together with the 95% confidence interval.

#### Further analyses

The patient's general condition (PGE) at Visit 1 and Visit 2, patient satisfaction at Visit 2 are categorical variables so they will be analysed as tabulations of frequencies. Change from Visit 1 to Visit 2 in the PF-10 score is a continuous outcome so it will be analysed with N / mean / SD / min / median / max.

The safety data will be reported according to local requirements. As similar studies will also be performed in other European countries, data pooling might be considered at the end.

#### 9.7.4 Handling of missing data

If less than half of the PF-10 questions are missing for a patient, the missing values will be replaced with the mean of the other values, then the PF-10 score will be calculated. If half or more than half of the PF-10 questions are missing, no score will be calculated and the PF-10 score will be marked as missing. No other missing data will be imputed. Every effort will be made to collect complete data at the specified time points.

Any removal from the analysis will be documented, stating the site and patient number as well as the reason for removal.

#### 9.8 QUALITY CONTROL

To improve and secure data quality, automatic data checks upon data entry will be done within the eCRF. In the eCRF, plausible ranges of values for numeric data entries as well as logical data entries and listings will be provided for each entry field. Based on this, checks on completeness and plausibility will be performed upon data entry in the eCRF.

Validity of data entry thus is ensured by integrated validation checks performed by the system, indicating missing or implausible entries to the document list or investigator. All corrections will be visible from the systems audit trail.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

No regular source data verification is planned in this study. However, in case of decreasing compliance (i.e. of missing data, data discrepancies, protocol violations, etc.) a for-cause audit or risk-based monitoring visit will be performed.

#### 9.9 LIMITATIONS OF THE RESEARCH METHODS

The intention of this NIS is to collect new data on the physical functioning and exercise capacity of COPD patients on treatment with Spiolto<sup>®</sup> Respirat<sup>®</sup> in a real world setting.

A NIS is the most suitable instrument for obtaining information about the use of medicines in everyday therapeutic practice and thus for investigating prospectively questions in everyday therapeutic practice.

Consecutive enrolment will be employed to minimize selection bias. The entry criteria are non-restrictive which will permit the enrolment of a broad patient population. The choice of treatment is at the discretion of the investigator.

Selection bias could occur at the site level and the patient level. To minimize the site level selection bias, the goal is to have participating centers that have access to all available treatment options which are approved for use in that country for the targeted COPD patients. To minimize selection bias at the patient level, consecutive enrolment is performed. Information bias will be minimized by the use of standard eCRF, questionnaire and physicians' training on the study protocol.

An additional limitation is that the physical functioning questionnaire (PF-10) is assessing 10 items of the full 36-Item Short Form Health Survey (SF-36).

The 7-item satisfaction scale, which is to be completed by the patient in order to measure satisfaction with Spiolto<sup>®</sup> Respimat<sup>®</sup> use, is a self-designed Boehringer-Ingelheim scale, without a public source or validation status.

#### 9.10 OTHER ASPECTS

#### 9.10.1 Informed Consent, Data Protection, Study Records

The study will be carried out in compliance with the protocol, the principles laid down in the Declaration of Helsinki, and as close as possible to the standards of the International Conference of Harmonisation (ICH) Tripartite Guideline for Good Clinical Practice (GCP), Guidelines for Good Epidemiological Practice (GEP) [R10-4560], Good Pharmacoepidemiology Practice (GPP) [R09-0182] and relevant BI Standard Operating Procedures (SOPs).

Standard medical care (prophylactic, diagnostic and therapeutic procedures) remains in the responsibility of the treating physician of the patient.

The investigator should inform the sponsor immediately of any urgent safety measures taken to protect the study subjects against any immediate hazard, and also of any serious breaches of the protocol/ICH GCP.

The rights of the investigator and of the sponsor with regard to publication of the results of this study are described in the investigator contract. As a general rule, no study results should be published prior to finalization of the Study Report.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Insurance Cover: The requirements for insurance depend on local law and legislations in the participating country. If required, the terms and conditions of the insurance cover are made available to the investigator and the patients, and the documentation must be archived in the Investigator Site File (ISF).

#### 9.10.1.1 Study Approval, Patient Information, and Informed Consent

This study will be initiated only after all required legal documentation has been reviewed and approved by the respective Independent Ethics Committee (IEC) and competent authority (CA) according to national and international regulations. The same applies for the implementation of changes introduced by amendments.

The NIS will be reviewed by the submitted to the competent Ethics Committee before it starts, as will any amendments to the observational plan. A copy of the opinion can be found in the appropriate section of the clinical trial master file.

In addition, every participating physician is to be advised by his/her ethics committee in accordance with the rules of professional conduct.

Prior to patient participation in the study, written informed consent must be obtained from each patient (or the patient's legally accepted representative). Each signature must be personally dated by each signatory and the informed consent and any additional patient-information form retained by the investigator as part of the study records. A signed copy of the informed consent and any additional patient information must be given to each patient or the patient's legally accepted representative.

The patient must be informed that his/her personal study-related data will be used by Boehringer Ingelheim in accordance with the local data protection law. The level of disclosure must also be explained to the patient.

The patient must be informed that his / her medical records may be examined by authorized monitors (CML/CRA) or Clinical Quality Assurance auditors appointed by Boehringer Ingelheim, by appropriate IEC members, and by inspectors from regulatory authorities.

The observing physician will keep the original documents in accordance with the legal storage period.

#### 9.10.1.2 Data Quality Assurance

A quality assurance audit/inspection of this study may be conducted by the sponsor or sponsor's designees or by IECs or by regulatory authorities. The quality assurance auditor will have access to all medical records, the investigator's study-related files and correspondence, and the informed consent documentation of this study.

#### 9.10.1.3 Records

Case Report Forms (eCRFs) for individual patients will be provided by the sponsor via remote data capture. All of the clinical data and site/investigator characteristics will be captured via a web-based Electronic Data Capturing system. The site staff will enter and edit the data via a secure network, with secure access features (username, password and secure identification – an electronic password system). A complete electronic audit trail will be maintained.

# BI Study Number 1237.45 c06524595-04 Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Patients must not be identified on the eCRF by name. Appropriately coded identification (i.e. Patient numbers) must be used.

All patient questionnaires will be paper-based and will be left at the site upon completion by the patient.

#### 9.10.1.3.1 Source Documents

Source documents provide evidence for the existence of the patient and substantiate the integrity of the data collected. Source documents are filed at the investigator's site.

Data entered in the eCRFs that are transcribed from source documents must be consistent with the source documents or the discrepancies must be explained. The investigator may need to request previous medical records or transfer records; also current medical records must be available.

For the eCRF, the following data must be derived from source documents:

- Patient demographics (age, gender, height, and weight);
- History of smoking
- Reported exacerbations
- Past COPD therapies (6 months before visit 1)
- Respirat® training (Yes/No)
- GOLD spirometric classification (1,2, 3, 4)
- GOLD patient groups (A, B, C, D)
- Concomitant diseases / Comorbidities
- Concomitant COPD and other relevant medication
- Breathlessness based on mMRC score
- Physical Functioning (PF-10) Questionnaire
- Patient Satisfaction Questionnaire
- Adverse Drug Reactions (ADR & SADR), fatal AEs, pregnancies
- Rational for Spiolto<sup>®</sup> Respimat<sup>®</sup> treatment discontinuation (if applicable)
- Details of treatment continuation / discontinuation

#### 9.10.1.3.2 Direct Access to Source Data and Documents

The investigator / institution will permit study-related monitoring, audits, IEC review and regulatory inspection, providing direct access to all related source data / documents. eCRFs and all source documents, including progress notes and copies of laboratory and medical test results must be available at all times for review by the sponsor's clinical study monitor, auditor and inspection by health authorities. The Clinical Research Associate (CRA) / on site monitor and auditor may review all eCRFs, and written informed consents. The accuracy of the data will be verified by reviewing the documents described in section 9.10.1.3.1.

#### 9.10.1.4 Statement of Confidentiality

Individual patient medical information obtained as a result of this study is considered confidential and disclosure to third parties is prohibited with the exceptions noted below. Patient confidentiality will be ensured by using patient identification code numbers.

## Boehringer Ingelheim  BI Study Number 1237.45


c06524595-04

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Data generated as a result of the study need to be available for inspection on request by the participating physicians, the sponsor's representatives, by the IEC and the regulatory authorities, i.e. the competent authority (CA).

## 9.10.1.5 Completion of Study

The EC/competent authority in each participating EU member state needs to be notified about the end of the trial (last patient/patient out, unless specified differently in <u>section 6</u> of the observational plan) or early termination of the trial.

#### 9.10.1.6 Protocol Violations

There are no protocol waivers. All protocol violations must be reported to the sponsor immediately.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 10. PROTECTION OF HUMAN SUBJECTS

Please refer to section 9.10.1

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

#### 11.1 DEFINITIONS OF ADVERSE EVENTS

#### Adverse event

An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (e.g. an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

#### Adverse drug reaction

An adverse drug reaction (ADR) is defined as a response to a medicinal product which is noxious and unintended. Response in this context means that a causal relationship between a medicinal product and an adverse event is at least a reasonable possibility. Adverse drug reactions may arise from use of the product within or outside the terms of the marketing authorization or from occupational exposure. Conditions of use outside the marketing authorization include off-label use, overdose, misuse, abuse and medication errors.

#### Serious adverse event

A serious adverse event is defined as any AE which

- results in death,
- is life-threatening,
- requires in-patient hospitalization, or
- prolongation of existing hospitalization,
- results in persistent or significant disability or incapacity, or
- is a congenital anomaly/birth defect

Life-threatening in this context refers to a reaction in which the patient was at risk of death at the time of the reaction; it does not refer to a reaction that hypothetically might have caused death if more severe.

Medical and scientific judgment should be exercised in deciding whether other situations should be considered serious reactions, such as important medical events that might not be immediately life threatening or result in death or hospitalization but might jeopardize the patient or might require intervention to prevent one of the other outcomes listed above.

Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization or development of dependency or abuse. Any suspected transmission via a medicinal product of an infectious agent is also considered a serious adverse reaction.

#### Adverse Event of Special Interest (AESI)

The term AESI relates to any specific AE that has been identified at the project level as being of particular concern for prospective safety monitoring and safety assessment within this

**BI Study Number 1237.45** 

c06524595-04

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

study, e.g. the potential for AEs based on knowledge from other compounds in the same class.

No AESIs have been defined for this study.

# 11.2 ADVERSE EVENT AND SERIOUS ADVERSE EVENT COLLECTION AND REPORTING

The investigator shall maintain and keep detailed records of all AEs in their patient files.

#### Collection of AEs

The study design is of non-interventional nature and the study is conducted within the conditions of the approved marketing authorisation. Sufficient data from controlled interventional trials are available to support the evidence on the safety and efficacy of the studied BI drug. For this reason the following AE collection and reporting requirements have been defined.

The following must be collected by the investigator in the eCRF from signing the informed consent onwards until the end of the study:

- all ADRs (serious and non-serious),
- all AEs with fatal outcome (serious adverse events),

Note\*: For all patients on these data must be recorded on the AE pages in the eCRF. The separate NIS (S)AE form must be used only when eCRF system is unavailable and must be forwarded to the local Pharmacovigilance fax as indicated in the form.

All ADRs, including those persisting after study completion must be followed up until they are resolved, have been sufficiently characterized, or no further information can be obtained.

The investigator carefully assesses whether an AE constitutes an ADR using the information below.

#### Causal relationship of adverse event

The definition of an adverse reaction implies at least a reasonable possibility of a causal relationship between a suspected medicinal product and an adverse event. An adverse reaction, in contrast to an adverse event, is characterized by the fact that a causal relationship between a medicinal product and an occurrence is suspected.

Medical judgment should be used to determine the relationship, considering all relevant factors, including pattern of reaction, temporal relationship, de-challenge or re-challenge, confounding factors such as concomitant medication, concomitant diseases and relevant history.

Arguments that may suggest a **reasonable causal relationship** could be:

- The event is **consistent with the known pharmacology** of the drug
- The event is known to be caused by **or attributed to the drug class**.
- A plausible time to onset of the event relative to the time of drug exposure.
- Evidence that the **event is reproducible** when the drug is re-introduced

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- **No medically sound alternative etiologies** that could explain the event (e.g. preexisting or concomitant diseases, or co-medications).
- The event is typically **drug-related and infrequent in the general population** not exposed to drugs (e.g. Stevens-Johnson syndrome).
- An indication of dose-response (i.e. greater effect size if the dose is increased, smaller effect size if dose is diminished).

Arguments that may suggest that there is **no reasonable possibility of a causal relationship** could be:

- No plausible time to onset of the event relative to the time of drug exposure is evident (e.g. pre-treatment cases, diagnosis of cancer or chronic disease within days/weeks of drug administration; an allergic reaction weeks after discontinuation of the drug concerned)
- Continuation of the event despite the withdrawal of the medication, taking into account the pharmacological properties of the compound (e.g. after 5 half-lives). Of note, this criterion may not be applicable to events whose time course is prolonged despite removing the original trigger.
- Additional arguments amongst those stated before, like alternative explanation (e.g. situations where other drugs or underlying diseases appear to provide a more likely explanation for the observed event than the drug concerned).
- Disappearance of the event even though the study drug treatment continues or remains unchanged.

#### Intensity of adverse event

The intensity of the AE should be judged based on the following:

Mild: Awareness of sign(s) or symptom(s) which is/are easily tolerated

Moderate: Enough discomfort to cause interference with usual activity

Severe: Incapacitating or causing inability to work or to perform usual activities

#### Pregnancy:

In rare cases, pregnancy might occur in this study. Once a subject has been enrolled into the study with Spiolto<sup>®</sup> Respimat<sup>®</sup>, the investigator must report any drug exposure during pregnancy, which occurred in a female subject or in a partner to a male subject, to the Sponsor by means of Part A of the Pregnancy Monitoring Form. The outcome of the pregnancy associated with the drug exposure during pregnancy must be followed up and reported by means of Part B of the Pregnancy Monitoring Form.

In the absence of a reportable AE, only the Pregnancy Monitoring Form must be completed, otherwise the NIS AE form is to be completed and forwarded (by fax) to the local Pharmacovigilance point of contact for each country within respective timelines.

#### Expedited Reporting of ADRs / Fatal AEs and Drug Exposure During Pregnancy

The following must be reported by the investigator on the NIS (S)AE Form from signing the informed consent onwards until the end of the study:

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 11.2:1 Reporting types and timelines

| Type of Report* | Timeline |
|---|---|
| All SADRs associated with Spiolto® Respimat® | immediately within 24 hours |
| All <b>AEs with fatal outcome</b> in patients exposed to Spiolto <sup>®</sup> Respimat <sup>®</sup> | immediately within 24 hours |
| All <b>non-serious ADRs</b> associated with Spiolto <sup>®</sup> Respimat <sup>®</sup> | 7 calendar days |
| All <b>pregnancy monitoring</b> forms associated with Spiolto <sup>®</sup> Respimat <sup>®</sup> | 7 calendar days |

The same timelines apply if follow-up information becomes available for the respective events. In specific occasions the Investigator could inform the Sponsor upfront via telephone. This does not replace the requirement to complete and fax/email the NIS (S)AE form.

#### Information required

For each reportable adverse event, the investigator should provide the information requested on the appropriate (e)CRF pages and the NIS (S)AE form.

#### Reporting of related Adverse Events associated with any other BI drug

The investigator is encouraged to report all adverse events related to any BI drug other than the Spiolto® Respimat® according to the local regulatory requirements for spontaneous AE reporting at the investigator's discretion by using the locally established routes and AE report forms. The term AE includes drug exposure during pregnancy, and, regardless of whether an AE occurred or not, any abuse, off-label use, misuse, medication error, occupational exposure, lack of effect, and unexpected benefit.

#### 11.3 REPORTING TO HEALTH AUTHORITIES

Adverse event reporting to regulatory agencies will be done by the Sponsor according to local and international regulatory requirements.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

Results of this non-interventional study will be disclosed on encepp.eu and clinicaltrials.gov and a study specific publication plan will be developed to describe planned publications.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 13. REFERENCES

(2006)

- 13.1 PUBLISHED REFERENCES P05-09483 Maltais F, Hamilton A, Marciniuk D, Hernandez P, Sciurba FC, Richter K, Kesten S, O'Donnell D Improvements in symptom-limited exercise performance over 8 h with once-daily tiotropium in patients with COPD. Chest 128 (3), 1168 - 1178 (2005) Guidelines for Good Pharmacoepidemiology Practices (GPP). R09-0182 Pharmacoepidemiology and Drug Safety 17, 200 - 208 (2008). Good Epidemiological Practice (GEP). IEA Guidelines for Proper Conduct of R10-4560 Epidemiological Reseach (2007). R13-3633 Troosters T1, Sciurba F, Battaglia S, Langer D, Valluri SR, Martino L, Benzo R. Andre D. Weisman I. Decramer M. Physical inactivity in patients with COPD, a controlled multi-center pilot-study. Respir Med. 2010 Jul;104(7):1005-11. doi: 10.1016/j.rmed.2010.01.012. Epub 2010 Feb 18 R15-5015 Claudio Tantucci, Denise Modina. Lung function decline in COPD. International Journal of COPD. 2012:7, 95-99. R15-4559 Katz P, Chen H, Omachi TA, Gregorich SE, Julian L, Cisternas M, Balmes J, Blanc PD Therole of physical inactivity in increasing disability among older adults with obstructive airway disease. J Cardiopulm Rehabil Prev 31 (3), 193 - 197 (2011) R15-4561 Maltais F, LeBlanc P, Simard C, Jobin J, Berube C, Bruneau J, Carrier L, Belleau R Skeletalmuscle adaptation to endurance training in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med 154, 442 -447 (1996) R15-4564 Garcia-Aymerich J, Lange P, Benet M, Schnohr P, Anto JM Regularphysical activity reduces hospital admission and mortality in chronic obstructive pulmonary disease: a population based cohort study. Thorax 61, 772 - 778
- P10-07776 Bouyssou T, Casarosa P, Naline E, Pestel S, Konetzki I, Devillier P, Schnapp A. Pharmacological characterization of olodaterol, a novel inhaled beta2-adrenoceptor agonist exerting a 24-hour-long duration of action in preclinical models. J Pharmacol Exp Ther 334 (1), 53 62 (2010)
- P10-09337 Bouyssou T, Schnapp A, Casarosa P, Pieper MP. Addition of the new oncedaily LABA BI 1744 to tiotropium results in superior bronchoprotection in pre-clinical models. ATS 2010, 106th Int Conf of the American Thoracic Society (ATS), New Orleans, 14 19 May 2010. Am J Respir Crit Care Med 181, A4445, Abstr (2010)

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- P10-14042 Maltais F, Beck E, Webster D, Maleki-Yazdi MR, Seibt JV, Arnoux A, Hamilton A. Four weeks once daily treatment with tiotropium + olodaterol (BI 1744) fixed dose combination compared with tiotropium in COPD patients. 20th Ann Cong of the European Respiratory Society (ERS), Barcelona, 18 22 Sep 2010. Eur Respir J 36 (Suppl 54), 1014S, Abstr 5557 (2010)
- P11-07720 Casarosa P, Kollak I, Kiechle T, Ostermann A, Schnapp A, Kiesling R, Pieper M, Sieger P, Gantner F. Functional and biochemical rationales for the 24-hour-long duration of action of olodaterol. J Pharmacol Exp Ther 337 (3), 600 609 (2011)
- P13-02357 Aalbers R, Maleki-Yazdi MR, Hamilton A, Waitere-Wijker S, Pivovarova A, Schmidt O, Bjermer L. Dose-finding study for tiotropium and olodaterol when administered in combination via the Respirat inhaler in patients with COPD. 22nd Ann Cong of the European Respiratory Society (ERS), Vienna, 1 5 Sep 2012. Eur Respir J 40 (Suppl 56), 525S 526S, Abstr P2882 (2012)
- P13-04267 Cooper CB, Celli BR, Jardim JR, Wise RA, Legg D, Guo J, Kesten S. Treadmill endurance during 2-year treatment with tiotropium in patients with COPD: a randomized trial. Chest 144 (2), 490 497 (2013)
- P13-05794 Tashkin DP, Ferguson GT. Combination bronchodilator therapy in the management of chronic obstructive pulmonary disease. Respir Res (Lond) 14, 49 (2013)
- P13-11341 Koch A, Paggiaro P, Hamilton A, Hart L, Korducki L, Salvo MC de, Pizzichini E. Symptomatic benefit of olodaterol QD delivered via Respimat vs placebo and formoterol BID in patients with COPD: combined analysis from two 48-week studies. 23rd Ann Cong of the European Respiratory Society (ERS), Barcelona, 7 11 Sep 2013
- P13-11345 Koch A, Pizzichini E, Hamilton A, Hart L, Korducki L, Salvo MC de, Paggiaro P. Lung function efficacy of olodaterol QD delivered via Respimat vs placebo and formoterol BID in patients with COPD: two 48-week studies. 23rd Ann Cong of the European Respiratory Society (ERS), Barcelona, 7 11 Sep 2013
- P13-11346 Ferguson G, Feldman G, Hofbauer P, Hamilton A, Allen L, Korducki L, Sachs P. Lung function efficacy of olodaterol QD delivered via Respirat in COPD patients: results from two 48-week studies. 23rd Ann Cong of the European Respiratory Society (ERS), Barcelona, 7 11 Sep 2013
- P13-11467 Lange P, Aumann JL, Derom E, Hamilton A, Tetzlaff K, Ting N, Noord JA van. The 24-h FEV1 time profile of olodaterol QD delivered via Respirat in COPD: results from two 6-week studies. 23rd Ann Cong of the European Respiratory Society (ERS), Barcelona, 7 11 Sep 2013
- P13-14109 Maltais F, Kirsten AM, Hamilton A, Sousa D de, Wang F, Decramer M. Evaluation of the effects of olodaterol on exercise endurance in patients with

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

COPD: results from two 6-week studies. Chest 2013, 79th Ann Mtg of the American College of Chest Physicians, Chicago, 26 - 31 Oct 2013. Chest 144 (4) (Suppl), 748A, Abstr (2013)

- P13-14112 Feldman G, Bernstein JA, Hamilton A, Nivens C, LaForce C. The 24-hour FEV1 time profile of olodaterol once daily (QD) via Respimat and formoterol twice daily (BID) via Aerolizer in patients with COPD: results from two 6-week studies. Chest 2013, 79th Ann Mtg of the American College of Chest Physicians, Chicago, 26 31 Oct 2013. Chest 144 (4) (Suppl), 749A, Abstr (2013)
- P14-01052 Global Initiative for Chronic Obstructive Lung Disease (GOLD). Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease (updated 2014). http://www.goldcopd.org/uploads/users/files/GOLD\_Report\_2014.pdf (access date: 22 January 2014); Global Initiative for Chronic Obstructive Lung Disease (GOLD) (2014)
- P14-12073 Bouyssou T, Casarosa P, Pieper M, Schnapp A, Gantner F. Synergistic bronchoprotective activity of the long-acting beta 2-agonist olodaterol with tiotropium (long-acting M3 antagonist) and ciclesonide (inhaled steroid) on the ovalbumin-induced bronchoconstriction in anaesthetized guinea pigs. ERJ September 1, 2011 vol. 38 no. Suppl 55 3451
- P13-14109 Maltais F, Kirsten AM, Hamilton A, Sousa D de, Wang F, Decramer M Evaluation of the effects of olodaterol on exercise endurance in patients with COPD: results from two 6-week studies. Chest 2013, 79th Ann Mtg of the American College of Chest Physicians, Chicago, 26 31 Oct 2013 Chest 144 (4) (Suppl), 748A, Abstr (2013)
- P15-03349 Buhl R, Maltais F, Abrahams R, Bjermer L, Derom E, Ferguson G, Flezar M, Hébert J, McGarvey L, Pizzichini E, Reid J, Veale A, Grönke L, Hamilton A, Korducki L, Tetzlaff K, Waitere-Wijker S, Watz H, Bateman E. Tiotropium and olodaterol fixed-dose combination versus mono-components in COPD (GOLD 2–4) Eur Respir J 2015; DOI: 10.1183/09031936.00136014
- P15-04531 Kai-Bichael Beeh, et al. The 24-h lung-function profile of once-daily tiotropium and olodaterol fixed-dose combination in chronic obstructive pulmonary disease. Elsevier Ltd, 2015. 1094-5539
- P94-1346 Bone R, et al. In chronic obstructive pulmonary disease, a combination of ipratropium and albuterol is more effective than either agent alone: an 85-day multicenter trial. Chest 105 (5), 1411 1419 (1994)

#### 13.2 UNPUBLISHED REFERENCES

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### ANNEX 1. LIST OF STAND-ALONE DOCUMENTS

The stand-alone documents for this non-interventional study are:

- Informed Consent Form
- Physicians' Global Evaluation (PGE)
- PF-10 Questionnaire based on SF-36
- Breathlessness Scale (mMRC)
- Patient Satisfaction Survey
- Statistical Epidemiological Analysis Plan (SEAP)
- Data Management Plan (DMP)
- Pregnancy Monitoring Form
- Serious Adverse Event Report in Non-Interventional Studies (NIS (S)AE Form)
- Publication Plan

All of the above documents will be archived in the Trial Master File in its original English master version.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## ANNEX 2. ENCEPP CHECKLIST FOR STUDY PROTOCOLS

Not applicable.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## **ANNEX 3. ADDITIONAL INFORMATION**

# Physical Functioning Questionnaire (PF-10) based on the 36-Item Short Form Survey.

| Please circle one number on each line. | | Yes,<br>Limited a<br>Lot | Yes,<br>Limited a<br>Little | No, Not limited at All |
|---|---|---|---|---|
| 1. | <b>Vigorous activities</b> , such as running, lifting heavy objects, participating in strenuous sports | [1] | [2] | [3] |
| 2. | Moderate activities, such as moving a table, pushing a vacuum cleaner, bowling, or playing golf | [1] | [2] | [3] |
| 3. | Lifting or carrying groceries | [1] | [2] | [3] |
| 4. | Climbing several flights of stairs | [1] | [2] | [3] |
| 5. | Climbing one flight of stairs | [1] | [2] | [3] |
| 6. | Bending, kneeling, or stooping | [1] | [2] | [3] |
| 7. | Walking more than a mile | [1] | [2] | [3] |
| 8. | Walking several blocks | [1] | [2] | [3] |
| 9. | Walking one block | [1] | [2] | [3] |
| 10. | Bathing or dressing yourself | [1] | [2] | [3] |

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## Modified Medical Research Council (mMRC) dyspnea (breathlessness) scale

## Please circle the number which best describes your grade of breathlessness.

| I only get breathless with strenuous exercise. | 0 |
|---|---|
| I get short of breath when hurrying on level ground or walking up a slight hill. | 1 |
| On level ground, I walk slower than people of the same age because of breathlessness, or have to stop for breath when walking at my own pace. | 2 |
| I stop for breath after walking about 100 yards or after a few minutes on level ground. | 3 |
| I am too breathless to leave the house or I am breathless when dressing. | 4 |

**BI Study Number 1237.45** 

c06524595-04

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **Patient Satisfaction Questionnaire**

Please circle the number which best describes your satisfaction with Spiolto<sup>®</sup> Respimat<sup>®</sup>.

What is your overall satisfaction with the Spiolto® Respimat® treatment?

1 2 3 4 5 6 7
very dissatisfied dissatisfied rather dissatisfied nor dissatisfied nor dissatisfied rather satisfied rather sa

How satisfied are your with inhaling from the Respimat® device (e.g. feeling of inhalation, ease of inhalation, speed of inhalation)?

1 2 3 4 5 6 7
very dissatisfied dissatisfied rather dissatisfied neither satisfied rather s

How satisfied are your with the handling of the Respirat® inhalation device?

1 2 3 4 5 6 7
very dissatisfied dissatisfied rather dissatisfied nor dissatisfied nor dissatisfied rather satisfied rather sa

BI Study Number 1237.45 c06524595-04

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## Physicians' Global Evaluation (PGE) to be used directly within the eCRF

General condition of the patient at the initial examination (Visit 1) Please mark with a cross as applicable

Poor Satisfactory Good Excellent

1 2 3 4 5 6 7 8

General condition of the patient after approximately 6 weeks of treatment (Visit 2) Please mark with a cross as applicable

Poor Satisfactory Good Excellent

1 2 3 4 5 6 7 8